CLINICAL TRIAL: NCT04305951
Title: Combining Acupuncture and Acupressure for Dementia Elderly: an Assessor-blinded, Randomized Controlled Trial
Brief Title: Combining Acupuncture and Acupressure for Dementia Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Prof. Zhang Zhang-Jin, Professor, Associate Director (Clinical Affairs), The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UW 19-821
Record Dates: First submitted 2020-03-10; First posted 2020-03-12 (Actual); Results first posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Dementia
Keywords: Dementia; Cognitive impairment; Elderly; Acupuncture; CAT; Acupressure; CAE
MeSH Terms: conditions — Dementia; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Routine care group (No Intervention): Subjects assigned to this group will continue their routine care without receiving any acupuncture and acupressure treatment during the study period. The routine care may include physiotherapy and intellectual activities. Post-trial treatment of either CAT, CAE, or CAT+CAE will be offered to serve as a compensation for their participation.
- CAT group (Experimental): Subjects assigned to comprehensive acupuncture therapy (CAT) group will receive CAT treatment in addition to routine care.
  Interventions: Procedure: Comprehensive acupuncture therapy (CAT)
- CAE group (Experimental): Subjects assigned to 'Comfy Acupressure for the Elderly (CAE)' group will receive CAE in addition to routine care.
  Interventions: Procedure: Comfy Acupressure for the Elderly (CAE)
- CAT + CAE group (Experimental): Subjects assigned to CAT+CAE group will receive CAT+CAE in addition to routine care.
  Interventions: Procedure: Comprehensive acupuncture therapy (CAT); Procedure: Comfy Acupressure for the Elderly (CAE)

INTERVENTIONS:
Procedure: Comprehensive acupuncture therapy (CAT) — CAT will be conducted for 2 sessions per week for 12 consecutive weeks.
  The following 14 body acupoints with only manual stimulation will be used: HT7 (Shenmen), LI4 (Hegu), TH5 (Waiguan), ST36 (Zusanli), ST40 (Fenglong) and SP6 (Sanyinjiao) in two sides, and CV12 (Zhongwan) and CV4 (Guanyuan) in midline. Electrical stimulation will be conducted on the following frontal acupoints: GV20 (Baihui), EX-HN3 (Yintang), GB15 (Toulinqi), GB8 (Shuaigu), EX-HN5 (Taiyang), and ST8 (Touwei) on two sides, and left and right EX-HN1 (Sishencong).
  Disposable acupuncture needles (0.25 mm in diameter and 25-40 mm in length) will be inserted at a depth of 10-30 mm perpendicularly or obliquely into acupoints. Manual manipulation will be carried out for all acupoints to evoke needling sensation. Electrical stimulation is additionally delivered on the 6 pairs of the frontal acupoints. Each session of treatment will last 30 minutes.
  Arms: CAT + CAE group; CAT group
Procedure: Comfy Acupressure for the Elderly (CAE) — CAE intervention will be conducted for 3 times per week for 12 consecutive weeks.
  CAE consists of 12 steps which need about 15 minutes to complete and mainly concentrates on the acupoints on face, head, neck, and shoulder. The detailed CAE Operation Guide will be provided for the provider and the video demonstration is accessible at https://www.youtube.com/watch?v=pAqNIZPKmnM.
  Arms: CAE group; CAT + CAE group

SUMMARY:
This is an assessor-blinded, randomized controlled trial. A total of 248 (anticipated) elderly people aged ≥65 years with a mild to moderate dementia will be recruited from local nursing and care homes. They will be randomly assigned to routine care, CAT, CAE, and CAT+CAE with n = 62 subjects in each group. Subjects assigned to CAT, CAE, and CAT+CAE will respectively receive 2 sessions of CAT, 3 sessions of CAE, and a combination of both per week for 12 weeks. The primary outcome is the baseline-to-endpoint change in score of the Montreal Cognitive Assessment (MoCA). Secondary outcomes include various domains of MoCA, functional independence, psychological well-being, sleep quality, and level of pain. A generalized linear mixed-effect model will be used to compare outcomes over time among the four groups.

DETAILED DESCRIPTION:
Currently, there are about 100,000 people aged 65 years and older who are suffering from clinically diagnosed dementia in Hong Kong (HK). With an ageing population, this number will increase to 280,000 by 2036. Most dementia elderly live in nursing homes and elderly daycare centers. Dementia is the major cause of disability and dependency in elderly people. It poses a significant burden on caregivers, families, and the public healthcare system. Patients with dementia not only have a wide range of cognitive impairment, but also develop a variety of frailty-related symptoms, mainly including physical and psychological frailty, such as musculoskeletal deterioration, neurological disorders, sleep, emotional, and even psychotic symptoms. The overall purpose of the management of dementia elderly is to reduce dementia- and frailty-caused adverse outcomes that increase disability, dependency, hospitalization, and long-term care admission. However, there is a dearth of effective interventions improving the quality of life of elderly with dementia. The development of holistic management strategies that not only prevent and slow cognitive deterioration, but also reduce various other symptoms is therefore highly desired.

Acupuncture has been widely used in the local clinical practice. Numerous studies have shown the benefits of acupuncture in reducing cognitive deterioration in patients with cognitive impairment and dementia and animal models. Acupuncture is also effective in improving physical disability, rigidity, gait, and postural balance in aging adults with stroke and Parkinson's disease. A large body of evidence further confirms the effectiveness of various acupuncture regimens in treating pain, fatigue, sleep disturbance, anxiety, and depression. On the other hand, it is well demonstrated that, as a convenient therapy, acupressure has particular benefits in alleviating sleep disturbance, anxiety, depression, and agitation in elderly with dementia. Acupressure also has positive effects on the recovery of motor function and daily activities of stroke patients. These studies suggest that acupuncture and acupressure could produce benefits for the elderly with dementia.

Most recently, we have completed three clinical trials that evaluated the efficacy of acupuncture treatment of vascular dementia; stroke-caused cognitive deterioration , and chemotherapy-induced cognitive impairment. All these trials have consistently revealed that acupuncture was effective in alleviating cognitive impairment. We also have shown the effectiveness of a caregiver-performed acupressure on the general quality of life in frail older people and self-administered acupressure for insomnia disorder. The caregiver-performed acupressure protocol is called 'Comfy Acupressure for the Elderly (CAE)' and demonstration video is accessible at https://www.youtube.com/watch?v=pAqNIZPKmnM. Furthermore, our several studies have confirmed the efficacy of acupuncture in improving major depression ; insomnia and anxiety, poststroke depression and movement disability. Meanwhile, we have developed a novel acupuncture mode called comprehensive acupuncture therapy (CAT) that consists of dense frontal acupoints with additional electrical stimulation and multiple body acupoints. The efficacy of CAT has been well proven in our previous studies.

The working hypothesis is that CAT and CAE are feasible, safe, and could produce better management outcomes than routine care in improving cognitive impairment, frailty-related disability and dependency as well as comorbid symptoms of aged people with dementia. The aims of this study are: (1) to determine whether the conditions of cognitive impairment in the treatment groups improve significantly when compared to control; (2) to determine whether other symptoms (e.g., functional independence, pain, depression, and sleep disorder) in the treatment groups improve more than in control; and (3) to investigate whether acupuncture or acupressure is safe for the elderly with cognitive impairment or dementia.

ELIGIBILITY:
Inclusion Criteria:

* have a clinical diagnosis of any type of dementia or met the criteria of major and mild neurocognitive disorder based on the Fifth Edition of the Diagnostic and Statistical Manual of Mental Disorders (DSM-5), and
* have mild to moderate dementia at a stage of 3-5 on the Global Deterioration Scale (GDS).

Exclusion Criteria:

* have of dementia with the stage below 3 or above 5 on the GDS;
* have severe skin lesions on acupuncture and acupressure areas;
* have significant bleeding tendency;
* have heart pacemaker or implantable cardioverter defibrillator;
* are currently receiving acupressure as a regular therapy;
* had a surgery on the head or neck;
* are currently receiving anti-coagulant treatment.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 236 (Actual)
Dates: Start 2021-10-05 (Actual); Primary Completion 2024-08-27 (Actual); Study Completion 2025-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zhang-Jin Zhang, MMed, PhD, Principal Investigator — School of Chinese Medicine, The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chan CWC, Chau PH, Leung AYM, Lo KC, Shi H, Yum TP, Lee YY, Li L. Acupressure for frail older people in community dwellings-a randomised controlled trial. Age Ageing. 2017 Nov 1;46(6):957-964. doi: 10.1093/ageing/afx050. PMID 28472415
- [Background] Chung KF, Yeung WF, Yu BY, Leung FC, Zhang SP, Zhang ZJ, Ng RM, Yiu GC. Acupuncture with or without combined auricular acupuncture for insomnia: a randomised, waitlist-controlled trial. Acupunct Med. 2018 Feb;36(1):2-13. doi: 10.1136/acupmed-2017-011371. Epub 2017 Dec 11. PMID 29229613
- [Background] Hmwe NTT, Browne G, Mollart L, Allanson V, Chan SW. An integrative review of acupressure interventions for older people: A focus on sleep quality, depression, anxiety, and agitation. Int J Geriatr Psychiatry. 2019 Mar;34(3):381-396. doi: 10.1002/gps.5031. Epub 2018 Dec 10. PMID 30430640
- [Background] Kwan RYC, Leung MCP, Lai CKY. A Randomized Controlled Trial Examining the Effect of Acupressure on Agitation and Salivary Cortisol in Nursing Home Residents with Dementia. Dement Geriatr Cogn Disord. 2017;44(1-2):92-104. doi: 10.1159/000478739. Epub 2017 Jul 29. PMID 28768251
- [Background] Man SC, Hung BH, Ng RM, Yu XC, Cheung H, Fung MP, Li LS, Leung KP, Leung KP, Tsang KW, Ziea E, Wong VT, Zhang ZJ. A pilot controlled trial of a combination of dense cranial electroacupuncture stimulation and body acupuncture for post-stroke depression. BMC Complement Altern Med. 2014 Jul 19;14:255. doi: 10.1186/1472-6882-14-255. PMID 25038733
- [Background] Margenfeld F, Klocke C, Joos S. Manual massage for persons living with dementia: A systematic review and meta-analysis. Int J Nurs Stud. 2019 Aug;96:132-142. doi: 10.1016/j.ijnurstu.2018.12.012. Epub 2019 Jan 4. PMID 30679034
- [Background] Qu SS, Huang Y, Zhang ZJ, Chen JQ, Lin RY, Wang CQ, Li GL, Wong HK, Zhao CH, Pan JY, Guo SC, Zhang YC. A 6-week randomized controlled trial with 4-week follow-up of acupuncture combined with paroxetine in patients with major depressive disorder. J Psychiatr Res. 2013 Jun;47(6):726-32. doi: 10.1016/j.jpsychires.2013.02.004. Epub 2013 Mar 14. PMID 23498306
- [Background] Simoncini M, Gatti A, Quirico PE, Balla S, Capellero B, Obialero R, D'Agostino S, Sandri N, Pernigotti LM. Acupressure in insomnia and other sleep disorders in elderly institutionalized patients suffering from Alzheimer's disease. Aging Clin Exp Res. 2015 Feb;27(1):37-42. doi: 10.1007/s40520-014-0244-9. Epub 2014 May 31. PMID 24878886
- [Background] Toosizadeh N, Lei H, Schwenk M, Sherman SJ, Sternberg E, Mohler J, Najafi B. Does integrative medicine enhance balance in aging adults? Proof of concept for the benefit of electroacupuncture therapy in Parkinson's disease. Gerontology. 2015;61(1):3-14. doi: 10.1159/000363442. Epub 2014 Oct 22. PMID 25341431
- [Background] Wang S, Yang H, Zhang J, Zhang B, Liu T, Gan L, Zheng J. Efficacy and safety assessment of acupuncture and nimodipine to treat mild cognitive impairment after cerebral infarction: a randomized controlled trial. BMC Complement Altern Med. 2016 Sep 13;16(1):361. doi: 10.1186/s12906-016-1337-0. PMID 27623621
- [Background] Wu YT, Ali GC, Guerchet M, Prina AM, Chan KY, Prince M, Brayne C. Prevalence of dementia in mainland China, Hong Kong and Taiwan: an updated systematic review and meta-analysis. Int J Epidemiol. 2018 Jun 1;47(3):709-719. doi: 10.1093/ije/dyy007. PMID 29444280
- [Background] Yang A, Wu HM, Tang JL, Xu L, Yang M, Liu GJ. Acupuncture for stroke rehabilitation. Cochrane Database Syst Rev. 2016 Aug 26;2016(8):CD004131. doi: 10.1002/14651858.CD004131.pub3. PMID 27562656
- [Background] Yang JW, Shi GX, Zhang S, Tu JF, Wang LQ, Yan CQ, Lin LL, Liu BZ, Wang J, Sun SF, Yang BF, Wu LY, Tan C, Chen S, Zhang ZJ, Fisher M, Liu CZ. Effectiveness of acupuncture for vascular cognitive impairment no dementia: a randomized controlled trial. Clin Rehabil. 2019 Apr;33(4):642-652. doi: 10.1177/0269215518819050. Epub 2019 Jan 23. PMID 30672317
- [Background] Yang MH, Lin LC, Wu SC, Chiu JH, Wang PN, Lin JG. Comparison of the efficacy of aroma-acupressure and aromatherapy for the treatment of dementia-associated agitation. BMC Complement Altern Med. 2015 Mar 29;15:93. doi: 10.1186/s12906-015-0612-9. PMID 25880034
- [Background] Yeung WF, Chung KF, Tso KC, Zhang SP, Zhang ZJ, Ho LM. Electroacupuncture for residual insomnia associated with major depressive disorder: a randomized controlled trial. Sleep. 2011 Jun 1;34(6):807-15. doi: 10.5665/SLEEP.1056. PMID 21629370
- [Background] Yeung WF, Ho FY, Chung KF, Zhang ZJ, Yu BY, Suen LK, Chan LY, Chen HY, Ho LM, Lao LX. Self-administered acupressure for insomnia disorder: a pilot randomized controlled trial. J Sleep Res. 2018 Apr;27(2):220-231. doi: 10.1111/jsr.12597. Epub 2017 Sep 8. PMID 28884877
- [Background] Yue S, Jiang X, Wong T. Effects of a nurse-led acupressure programme for stroke patients in China. J Clin Nurs. 2013 Apr;22(7-8):1182-8. doi: 10.1111/j.1365-2702.2012.04127.x. Epub 2012 Jul 17. PMID 22805254
- [Background] Zhang ZJ, Ng R, Man SC, Li TY, Wong W, Tan QR, Wong HK, Chung KF, Wong MT, Tsang WK, Yip KC, Ziea E, Wong VT. Dense cranial electroacupuncture stimulation for major depressive disorder--a single-blind, randomized, controlled study. PLoS One. 2012;7(1):e29651. doi: 10.1371/journal.pone.0029651. Epub 2012 Jan 6. PMID 22238631
- [Background] Zhang ZJ, Wang XM, McAlonan GM. Neural acupuncture unit: a new concept for interpreting effects and mechanisms of acupuncture. Evid Based Complement Alternat Med. 2012;2012:429412. doi: 10.1155/2012/429412. Epub 2012 Mar 8. PMID 22474503

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment and treatment started in October 2021 and ended in August 2024. Elderly people with cognitive impairment or dementia of any type were recruited in 19 local elderly care homes, with 6 in Hong Kong Island, 9 in Kowloon and 4 in New Territories.
Period: Overall Study
Arm/Group | Routine Care Group | CAT Group | CAE Group | CAT + CAE Group
Started | 59 | 59 | 59 | 59
Completed | 55 | 46 | 51 | 49
Not Completed | 4 | 13 | 8 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Routine Care Group | CAT Group | CAE Group | CAT + CAE Group | Total
Number analyzed (Participants) | 59 | 59 | 59 | 59 | 236
Age, Continuous [Mean (Standard Deviation); unit: year] | 85.3 (7.2) | 82.6 (8.8) | 84.8 (8.7) | 84.6 (8.6) | 84.3 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 30 | 35 | 31 | 137
  Male | 18 | 29 | 24 | 28 | 99
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
MoCA [Mean (Standard Deviation); unit: score] | 8.8 (5.9) | 10.5 (7.3) | 10.9 (7.3) | 10.1 (6.3) | 10.1 (6.7)

OUTCOME MEASURES:

1. Primary Outcome: Changes in the Montreal Cognitive Assessment Score
Description: Severity of dementia is primarily measured using Montreal Cognitive Assessment (MoCA) and its overall score ranges from 0 to 30. A higher score indicates better cognition. Assessments will be conducted at baseline and once every six weeks thereafter.
Time Frame: Baseline, 6 week, 12 week
Population: The efficacy was analyzed in the intention-to-treat population, defined as participants who have been randomized.
Measure: Mean (95% Confidence Interval); unit: score
Arm/Group | Routine Care Group | CAT Group | CAE Group | CAT + CAE Group
Number analyzed (Participants) | 59 | 59 | 59 | 59
score
  Week 6 | 0.14 [-0.75 to 1.02] | 0.70 [-0.18 to 1.59] | 1.06 [0.13 to 1.99] | 0.44 [-0.37 to 1.25]
  Week 12 | -0.25 [-1.11 to 0.62] | 0.60 [-0.28 to 1.49] | 1.33 [0.40 to 2.26] | 0.40 [-0.44 to 1.23]

2. Secondary Outcome: Change in the Digit Span Forward
Description: Severity of dementia is measured using Digit Span Forward and its overall score ranges from 0 to 14. A higher score indicates better cognition. Assessments will be conducted at baseline and once every six weeks thereafter.
Time Frame: Baseline, 6 week, 12 week
Population: The efficacy was analyzed in the intention-to-treat population, defined as participants who have been randomized.
Measure: Mean (95% Confidence Interval); unit: score
Arm/Group | Routine Care Group | CAT Group | CAE Group | CAT + CAE Group
Number analyzed (Participants) | 59 | 59 | 59 | 59
score
  Week 6 | 0.04 [-1.01 to 1.09] | -0.15 [-0.97 to 0.67] | 0.01 [-0.68 to 0.70] | 0.37 [-0.28 to 1.01]
  Week 12 | -1.59 [-2.61 to -0.56] | -0.61 [-1.43 to 0.21] | -0.01 [-0.71 to 0.68] | 0.30 [-0.37 to 0.97]

3. Secondary Outcome: Change in the Digit Span Reverse
Description: Severity of dementia is measured using Digit Span Reverse and its overall score ranges from 0 to 14. A higher score indicates better cognition. Assessments will be conducted at baseline and once every six weeks thereafter.
Time Frame: Baseline, 6 week, 12 week
Population: The efficacy was analyzed in the intention-to-treat population, defined as participants who have been randomized.
Measure: Mean (95% Confidence Interval); unit: score
Arm/Group | Routine Care Group | CAT Group | CAE Group | CAT + CAE Group
Number analyzed (Participants) | 59 | 59 | 59 | 59
score
  Week 6 | -0.04 [-0.53 to 0.44] | -0.43 [-0.92 to 0.07] | 0.10 [-0.36 to 0.57] | 0.15 [-0.35 to 0.65]
  Week 12 | -0.23 [-0.70 to 0.25] | 0.02 [-0.48 to 0.51] | 0.47 [0.00 to 0.94] | 0.23 [-0.28 to 0.74]

4. Secondary Outcome: Changes in the Modified Bathel Index Score
Description: Functional independence is measured using Modified Bathel Index (MBI) and its overall score ranges from 10 to 50. A higher score indicates better functional independence. Assessments will be conducted at baseline and once every six weeks thereafter.
Time Frame: Baseline, 6 week, 12 week
Population: The efficacy was analyzed in the intention-to-treat population, defined as participants who have been randomized.
Measure: Mean (95% Confidence Interval); unit: score
Arm/Group | Routine Care Group | CAT Group | CAE Group | CAT + CAE Group
Number analyzed (Participants) | 59 | 59 | 59 | 59
score
  Week 6 | 0.82 [-1.33 to 2.96] | 1.97 [-0.50 to 4.43] | 0.94 [-0.61 to 2.49] | 0.68 [-1.12 to 2.48]
  Week 12 | -0.93 [-3.04 to 1.17] | 3.11 [0.63 to 5.59] | 0.57 [-1.00 to 2.13] | 1.82 [-0.02 to 3.67]

5. Secondary Outcome: Changes in the Visual Analogue Scale Score
Description: Pain is evaluated using visual analogue scale (VAS) and its overall score ranges from 0 to 10. A higher score indicates greater severity. Assessments will be conducted at baseline and once every six weeks thereafter.
Time Frame: Baseline, 6 week, 12 week
Population: The efficacy was analyzed in the intention-to-treat population, defined as participants who have been randomized.
Measure: Mean (95% Confidence Interval); unit: score
Arm/Group | Routine Care Group | CAT Group | CAE Group | CAT + CAE Group
Number analyzed (Participants) | 59 | 59 | 59 | 59
score
  Week 6 | 0.11 [-0.60 to 0.81] | -0.43 [-1.09 to 0.23] | 0.01 [-0.65 to 0.67] | -0.57 [-1.20 to 0.06]
  Week 12 | -0.18 [-0.87 to 0.51] | -0.23 [-0.90 to 0.44] | -0.49 [-1.17 to 0.18] | -0.32 [-0.97 to 0.33]

6. Secondary Outcome: Changes in the Geriatric Depression Scale Score
Description: Depressive symptoms are measured using the 15-item Geriatric Depression Scale (GDS-15) and its overall score ranges from 0 to 15. A higher score indicates greater severity. Assessments will be conducted at baseline and once every six weeks thereafter.
Time Frame: Baseline, 6 week, 12 week
Population: The efficacy was analyzed in the intention-to-treat population, defined as participants who have been randomized.
Measure: Mean (95% Confidence Interval); unit: score
Arm/Group | Routine Care Group | CAT Group | CAE Group | CAT + CAE Group
Number analyzed (Participants) | 59 | 59 | 59 | 59
score
  Week 6 | -0.49 [-1.70 to 0.71] | -0.67 [-1.73 to 0.40] | -1.23 [-2.32 to -0.13] | -0.62 [-1.53 to 0.30]
  Week 12 | -1.47 [-2.68 to -0.26] | -0.39 [-1.45 to 0.66] | -1.85 [-2.99 to -0.72] | -0.75 [-1.67 to 0.18]

7. Secondary Outcome: Changes in the Insomnia Severity Index Score
Description: Sleep parameters are measured using Insomnia Severity Index (ISI) and its overall score ranges from 0 to 28. A higher score indicates more acute sleep disturbances. Assessments will be conducted at baseline and once every six weeks thereafter.
Time Frame: Baseline, 6 week, 12 week
Population: The efficacy was analyzed in the intention-to-treat population, defined as participants who have been randomized.
Measure: Mean (95% Confidence Interval); unit: score
Arm/Group | Routine Care Group | CAT Group | CAE Group | CAT + CAE Group
Number analyzed (Participants) | 59 | 59 | 59 | 59
score
  Week 6 | -0.12 [-1.71 to 1.48] | -0.45 [-1.72 to 0.83] | -0.38 [-1.91 to 1.15] | -0.50 [-1.57 to 0.57]
  Week 12 | -0.67 [-2.26 to 0.93] | -1.26 [-2.56 to 0.05] | -1.46 [-3.03 to 0.12] | -0.84 [-1.95 to 0.28]

ADVERSE EVENTS:
Time Frame: from enrollment until end of follow-up, up to 12 weeks
Arm/Group | Routine Care Group | CAT Group | CAE Group | CAT + CAE Group
All-Cause Mortality (participants affected / at risk) | 0/59 | 2/59 | 0/59 | 1/59
Serious Adverse Events (participants affected / at risk) | 3/59 | 5/59 | 6/59 | 3/59
Other Adverse Events (participants affected / at risk) | 1/59 | 15/59 | 1/59 | 15/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Routine Care Group (N=59) | CAT Group (N=59) | CAE Group (N=59) | CAT + CAE Group (N=59)
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0
COVID-19 infection (Infections and infestations) | 1 | 0 | 1 | 0
Patent foramen ovale-associated platypnea-orthodeoxia syndrome (Cardiac disorders) | 1 | 0 | 0 | 0
Diabetes (Endocrine disorders) | 0 | 1 | 0 | 0
Epilepsy (Nervous system disorders) | 0 | 1 | 0 | 0
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Hematuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Fall (General disorders) | 0 | 0 | 1 | 2
Diarrhea (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Fatigue (Investigations) | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 1 | 0
Heart failure (Cardiac disorders) | 0 | 2 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Routine Care Group (N=59) | CAT Group (N=59) | CAE Group (N=59) | CAT + CAE Group (N=59)
Bleeding at the site of needling (General disorders) | 0 | 7 | 0 | 4
Fall (General disorders) | 1 | 3 | 0 | 0
Fever (Infections and infestations) | 0 | 1 | 0 | 3
Hematoma around the site of needling (General disorders) | 0 | 4 | 0 | 5
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-08-21): https://cdn.clinicaltrials.gov/large-docs/51/NCT04305951/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-21): https://cdn.clinicaltrials.gov/large-docs/51/NCT04305951/SAP_001.pdf